CLINICAL TRIAL: NCT06064812
Title: A Phase I/II, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Efficacy of FWD1802in Patients With ER+/HER2- Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: A Phase I/II Study of FWD1802 in Patients With ER+/HER2- Advanced BC.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Forward Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FWD1802-001C
Record Dates: First submitted 2023-09-20; First posted 2023-10-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Breast Cancer; Locally Advanced Breast Cancer; Breast Cancer Stage IV; ER+/HER2- Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I Study Part A: Dose Escalation. (Experimental): Part A study will be conducted in subjects diagnosed with ER+/HER2- unresectable locally advanced or metastatic breast cancer. A maximum of 27 subjects will be enrolled. They will be sequentially allocated to 5 planned dose cohorts: 25 mg, 75 mg, 150 mg, 300 mg and 450 mg. Subjects enrolled will be orally administered a single dose of FWD1802 Tablet on C0D1, followed by a 3-day observation period. Starting on C1D1, FWD1802 Tablet will be orally administered continuously QD for 28 consecutive days of each cycle. The DLT observation period is set as 32 days(C0D1-C1D28). The second cycle and subsequent cycles will last for 28 days per cycle. The patients will continue to receive the study treatment until PD, death, unacceptable toxicity, withdrawal of informed consent, or other reasons to discontinue study treatment occurs, whichever comes first.
  Interventions: Drug: FWD1802
- Phase I Study Part B - Dose Expansion. (Experimental): Part B will be conducted based on the dose-escalation results from Part A (comprehensive safety, PK, PD, and other data), selecting 2 to 4 dose cohorts for further exploration of the PK characteristics and RP2D of FWD1802. Each dose cohort will be expanded to include a maximum of 10 subjects (this total includes subjects from the corresponding dose cohort in Part A).
  The doses selected for Part B must be within the dose levels already explored and confirmed as safe to ensure that all doses in Part B fall within a known safety range. The SMC will decide on the 2 to 4 doses for expansion, which may include doses already confirmed as safe in Part A or new doses within the established safe range.
  The timing for initiating Part B will be jointly determined by the SMC and the sponsor based on the information already obtained from Part A. Part B may commence concurrently with the dose-escalation phase. The 2 to 4 dose cohorts in Part B may be conducted simultaneously or sequentially.
  Interventions: Drug: FWD1802
- Phase II Study - Dose Expansion in ER+/HER2- Subjects with ESR1 Mutations. (Experimental): The dose expansion study will be conducted in approximately 60 subjects diagnosed with ER+/HER2- locally advanced or metastatic breast cancer harboring ESR1 mutations, to evaluate the efficacy, safety and PK of FWD1802 at the recommended 1 to 2 dose level(s).
  The specific number of subjects, dosage(s), and dosing regimen in the dose expansion study will be comprehensively determined by the SMC based on the results from the Phase I, Part A study.
  Subjects will undergo ctDNA testing before treatment initiation, on Cycle 1 Day 15 (C1D15), on Cycle 2 Day 1 (C2D1), after disease progression, and when deemed necessary based on the subject's therapeutic response, to determine the baseline mutation sites, types, and frequencies of ESR1 and/or other breast cancer-related genes.
  Interventions: Drug: FWD1802

INTERVENTIONS:
Drug: FWD1802 — Eligible subjects will receive FWD1802 treatment according to their assigned dose cohort.
  Dose Escalation Phase:
  This phase is divided into a Single-Agent Lead-in Period (C0) and a Multiple-Dosing Period (C1). During the single-agent lead-in period, subjects will receive one dose on Day 1, followed by a 6-day dosing pause. In the multiple-dosing period, subjects will be administered FWD1802 once daily.
  Dose Expansion Phase:
  Subjects will receive FWD1802 once daily. Each 4-week period constitutes one treatment cycle. Treatment will continue for up to 2 years or until one of the following events occurs (whichever comes first): disease progression, intolerable toxicity, withdrawal of informed consent, loss to follow-up, initiation of new anti-cancer therapy, or death. Patients who remain in the study at the end of the 2-year treatment period and continue to derive clinical benefit may, upon agreement between the investigator and the sponsor, have the option to continue treatment.

SUMMARY:
A Phase I/II, Open-label study to assess the safety, tolerability, pharmacokinetic, and antitumor efficacy of FWD1802 monotherapy in patients with ER+/HER2- unresectable locally advanced or metastatic breast cancer. This clinical trial aims to explore the role of FWD1802 in the ER+/HER2- advanced breast cancer patient population. The primary objectives are to address the following questions:

Phase I Study:

Determine the Recommended Phase II Dose (RP2D) and/or Maximum Tolerated Dose (MTD) of FWD1802 in patients with ER-positive, HER2-negative locally advanced or metastatic breast cancer.

Phase II Study:

To evaluate the efficacy of FWD1802 at the RP2D in patients with ESR1-mutated ER-positive/HER2-negative locally advanced or metastatic breast cancer, using objective response rate (ORR) as the efficacy endpoint.

DETAILED DESCRIPTION:
This is a phase I/II, multicenter, open-label, first-in-human study of FWD1802 in patients with locally advanced or metastatic breast cancer that is estrogen receptor (ER)-positive/human epidermal growth factor receptor 2 (HER2)-negative (Phase II: restricted to patients with ESR1-mutated). It consists of three parts: the FWD1802 dose-escalation phase (Phase I Part A), the FWD1802 dose-expansion phase (Phase I Part B), and the dose-expansion study of FWD1802 in patients with ESR1 mutations (Phase II study).

Each study phase includes a screening period (up to 4 weeks), a treatment period (maximum treatment duration of 2 years; continuation beyond 2 years is permitted if the investigator judges the subject is still benefiting, with agreement from both the investigator and sponsor), and a follow-up period. The Phase II study includes a pre-screening period; patients with unknown mutation status may undergo testing that includes ESR1 mutation status prior to the screening period.

Phase I Part A is the FWD1802 dose-escalation study: A dose-escalation trial using a combination of an "accelerated titration" design and a "3+3" design is planned, with a maximum of 27 subjects to be enrolled. The Safety Monitoring Committee (SMC) will evaluate pharmacokinetic (PK), pharmacodynamic (PD), efficacy, and safety data to guide the determination of potentially effective doses for Part B and the Phase II study.

Phase I Part B is the FWD1802 dose-expansion study: Based on safety, PK, PD, and other data obtained from Part A, 2 to 4 dose cohorts will be selected for further exploration of FWD1802's PK profile and the recommended phase 2 dose (RP2D). Each dose cohort will be expanded to include up to 10 subjects (including subjects from the corresponding dose cohort in Part A). The SMC will decide which dose cohorts to expand and the timing of expansion based on information obtained from Part A. Dose expansion may proceed concurrently with the dose-escalation phase, within dose ranges already confirmed as safe by the SMC.

The Phase II study is cohort expansion study targeting the population with ESR1 mutations: Enrolled subjects will have ER-positive, HER2-negative breast cancer with ESR1 mutations. One to two dose levels will be selected for exploration, with each dose level enrolling no more than 30 subjects, for a maximum total enrollment of 60 subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for enrollment in this clinical study:

1. Voluntarily participate in the clinical trial and sign the informed consent form.
2. Female, aged ≥18 years.
3. Able to provide blood samples for central laboratory testing of ESR1 mutation status and other biomarker assessments. Phase I Study: ESR1 mutation status will be tested retrospectively. Phase II Study: Only subjects with confirmed ESR1 mutations will be enrolled (see Appendix 5 for details).
4. Histologically or cytologically confirmed locally advanced or metastatic breast cancer that is ER-positive and HER2-negative.

   Criteria for ER positivity: Immunohistochemistry staining shows nuclear staining in ≥10% of tumor cells.

   Criteria for HER2 negativity: Immunohistochemistry staining intensity is 0 or 1+; if the intensity is 2+, it must be confirmed negative by in situ hybridization.
5. Confirmed in menopause and not caused by ovarian function suppression drugs, must meet one of the following criteria:

   Previous bilateral oophorectomy. Age ≥ 60 years.

   Age < 60 years (subdivided into the following conditions):
   1. Never received chemotherapy, ovarian function inhibitors, or SERM drugs (tamoxifen, toremifene), with amenorrhea ≥12 months, and E2 and FSH levels in the postmenopausal range.
   2. Received chemotherapy resulting in chemotherapy-induced amenorrhea ≥12 months, with E2 and FSH levels in the postmenopausal range.
   3. Using SERM drugs (tamoxifen, toremifene), with E2 and FSH levels in the postmenopausal range.
6. Premenopausal or perimenopausal female subjects must agree to receive and maintain treatment with ovarian function suppression (LHRH agonists) during the study treatment period (ovarian function suppression treatment must be initiated at least 14 days before the first dose of study drug).
7. Prior treatment history must meet the following requirements:

   1. Disease progression during or intolerance to standard therapy, or unsuitability for standard therapy.
   2. Previous adjuvant endocrine therapy for at least 2 years, with recurrence during treatment or within 1 year after completion; OR at least one line of endocrine therapy for the advanced stage, with progression after at least 6 months of maintenance therapy on any line of advanced endocrine therapy (no limit on the number of endocrine therapy lines).
   3. Previous chemotherapy for the advanced stage is ≤ 2 lines.
   4. Prior use of fulvestrant, with an interval of at least 6 weeks between the last dose of fulvestrant and the first dose in this study.
   5. An interval of at least 6 weeks is required between the last dose of prior tamoxifen and the first dose in this study.
   6. Previous treatment with CDK4/6 inhibitors is ≤ 1 line.
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 (see Appendix 1 for details).
9. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Tumor lesions that have previously received radiotherapy or other local-regional treatment can only be considered measurable lesions if disease progression is confirmed.
10. Expected survival ≥ 3 months.
11. Subjects must have adequate organ and bone marrow function at screening (no blood transfusion, human albumin administration, or use of hematopoietic growth factors within 7 days prior to screening tests), defined as follows:

    1. Complete Blood Count:

       Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L. White blood cell count (WBC) ≥ 3.0 × 10⁹/L and ≤ 15 × 10⁹/L. Platelet count (PLT) ≥ 100 × 10⁹/L. Hemoglobin (HGB) ≥ 100 g/L.
    2. Liver Function:

       Serum total bilirubin (TBIL) ≤ 1.5 × ULN. For subjects without liver metastases: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN.

       For subjects with liver metastases: ALT and AST ≤ 5 × ULN.
    3. Renal Function:

       Serum creatinine (Scr) ≤ 1.5 × ULN OR creatinine clearance (Clcr) calculated by the Cockcroft-Gault method ≥ 50 mL/min.
    4. Coagulation Function:

       Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

       International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN (for subjects on anticoagulant therapy, values should be within the therapeutic range):
       1. For patients receiving warfarin, INR must be stable between 2.0 and 3.0.
       2. For patients receiving heparin, APTT should be between 1.5 and 2.5 × ULN (or returned to the value prior to starting heparin therapy).
       3. For prosthetic heart valves requiring anticoagulation, a stable INR between 2.5 and 3.5 is allowed.
    5. Cardiac Function:

    Left ventricular ejection fraction (LVEF) > 50% as shown by echocardiography.
12. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose and must be non-lactating. Women of childbearing potential must agree to use effective contraceptive methods from the time of signing the informed consent form until 6 months after the last dose of the study drug. Effective methods include double barrier methods, condoms, oral or injectable contraceptives, intrauterine devices, etc. All female subjects will be considered of childbearing potential unless they are naturally postmenopausal, have undergone artificial menopause, or have undergone sterilization (e.g., hysterectomy, bilateral salpingo-oophorectomy).

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Leptomeningeal metastases, carcinomatous meningitis, spinal cord compression, or symptomatic or clinically unstable central nervous system (CNS) metastases.
2. History of ongoing gastrointestinal diseases or other malabsorptive conditions that may impact the absorption of orally administered study drugs, including but not limited to:

   1. Inability to swallow oral medications.
   2. Requirement for intravenous nutrition.
   3. Prior surgery affecting absorption, including total/partial gastrectomy.
   4. Crohn's disease, ulcerative colitis.
   5. Treatment for active peptic ulcer disease within 6 months prior to the first dose.
   6. Malabsorption syndrome, or uncontrolled nausea, vomiting, or diarrhea.
3. Patients with symptomatic visceral metastases, or those with clinically significant and unstable pleural, peritoneal, pericardial effusions, or pulmonary lymphangitic carcinomatosis. Patients who have received intracavitary infusion therapy or drainage/paracentesis may be enrolled 14 days or more after the effusion has stabilized. Other conditions deemed by the investigator as unsuitable for endocrine therapy.
4. Prior treatments do not meet the following washout periods:

   1. Use of other investigational drugs or devices within 4 weeks prior to the first dose.
   2. Treatment with CDK4/6 inhibitors or mTOR inhibitors within 2 weeks, or other targeted therapies, chemotherapy, or immunotherapy within 4 weeks prior to the first dose.
   3. Radiotherapy, endocrine drugs, or traditional Chinese medicines with anti-tumor indications within 2 weeks prior to the first dose (washout periods for fulvestrant and tamoxifen refer to Inclusion Criterion 7).
   4. Treatment with mitomycin or nitrosoureas within 6 weeks prior to the first dose.
   5. Use of drugs or herbal supplements known to be moderate/strong inhibitors or inducers of CYP3A4 within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose (see Appendix 4).
   6. Use of drugs that inhibit gastric acid production within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose (see Appendix 4).
   7. Use of drugs that are P-glycoprotein (P-gp) inhibitors within 2 weeks or 5 half-lives (whichever is longer) prior to the first dose (see Appendix 4).
5. Toxicities from prior anti-tumor therapy have not recovered to Grade ≤1 (except for alopecia, and chemotherapy-induced peripheral neuropathy ≤ Grade 2).
6. Major surgical procedure (excluding biopsy) within 4 weeks prior to the first dose of study drug, or incomplete healing of surgical incision.
7. Known other active malignancy within the past 5 years (except for cured basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, papillary thyroid carcinoma, or ductal carcinoma in situ of the breast).
8. History of interstitial lung disease, drug-induced interstitial lung disease, or any evidence of active pneumonitis on chest CT scan within 4 weeks prior to the first dose of study drug.
9. Poorly controlled hypertension despite antihypertensive therapy (systolic blood pressure >150 mmHg or diastolic blood pressure >95 mmHg).
10. Active hepatitis B (defined as HBsAg positive and HBV DNA >500 IU/mL or >2000 copies/mL, or HBV DNA above the lower limit of detection if the local lower limit is >500 IU/mL or >2000 copies/mL); hepatitis C virus (HCV) infection (defined as HCV antibody positive and HCV-RNA positive or HCV-RNA above the lower limit of detection at the local site).

    Known HIV infection or history of acquired immunodeficiency syndrome (AIDS); active tuberculosis; active syphilis infection.
11. Any severe infection requiring systemic antibiotics within 14 days prior to dosing, or active infection requiring systemic treatment.
12. Arterial or venous thrombotic events within 6 months, including cerebrovascular accident (e.g., transient ischemic attack, cerebral hemorrhage, etc.), deep vein thrombosis, or pulmonary embolism.
13. History of active cardiac disease or cardiac dysfunction, including any of the following:

    1. Idiopathic symptomatic bradycardia within 2 years prior to screening, or resting heart rate <50 bpm at screening.
    2. History of angina or symptomatic coronary artery disease within 1 year prior to screening.
    3. History of congestive heart failure (NYHA Class ≥3), cardiomyopathy, or myocardial ischemia requiring long-term medication for control.
    4. Acute myocardial infarction event within 6 months prior to screening.
    5. History of ventricular arrhythmia, or any supraventricular arrhythmia ≥ Grade 2 requiring treatment or intervention within 1 year prior to screening, or presence of risk factors for ventricular arrhythmias.
    6. Any factors that increase the risk of QTc prolongation or arrhythmic events, such as symptomatic heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under age 40 in a first-degree relative. Hypertrophic cardiomyopathy and clinically significant valvular stenosis.
    7. Poorly controlled atrial fibrillation, history of coronary/peripheral artery bypass graft within the past 6 months, or cerebrovascular symptoms including transient ischemic attack.
    8. QTcF (Fridericia's correction) > 470 ms on ECG.
    9. Presence of ECG abnormalities considered clinically significant by the investigator, including complete left bundle branch block, second- or third-degree heart block, or sick sinus syndrome.
14. History of severe allergic reactions to the study drug(s) or excipients used in the protocol.
15. Prior use of any selective estrogen receptor degrader (other than fulvestrant) or investigational drugs inhibiting the ER signaling pathway.
16. Patients with active or chronic corneal disease, other active eye disease requiring ongoing treatment, or any clinically significant corneal disease for which drug-induced keratopathy cannot be adequately monitored.
17. History of drug abuse, alcohol abuse, or substance abuse.
18. Use of live or attenuated live vaccines within 4 weeks prior to the first dose of study drug. Use of immunomodulatory drugs, including but not limited to thymosin, interleukin-2, interferon, etc., within 14 days prior to the first dose of study drug. History of allogeneic organ transplantation, allogeneic peripheral hematopoietic stem cell transplantation, or bone marrow transplantation.
19. Conditions deemed by the investigator as unsuitable for participation in this study, including but not limited to a clear history of neurological disorders such as epilepsy or dementia, poor compliance, or any other circumstances the investigator believes may render the subject unsuitable for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female
Enrollment: 99 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Phase I Study | Approximately 2 years
  Dose-Limiting Toxicity (DLT) Maximum Tolerated Dose (MTD) Recommended Phase II Dose (RP2D)
Phase II Study | Approximately 2 years
  Objective Response Rate (ORR) as assessed by the investigator per RECIST v1.1

SECONDARY OUTCOMES:
Phase I Study | Approximately 2 years]
  Safety Endpoints: Laboratory parameters, 12-lead electrocardiogram (ECG), vital signs, treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). The incidence of AEs/SAEs, their severity and relationship to the study drug will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
  Pharmacokinetic Endpoints: PK parameters of FWD1802 including time to maximum plasma concentration (Tmax), maximum plasma concentration (Cmax), area under the plasma concentration-time curve (AUC, including AUC0-t and AUC0-∞), and terminal elimination half-life (T1/2).
  Efficacy Endpoints:
  ORR, Clinical Benefit Rate (CBR), Duration of Response (DoR), Disease Control Rate (DCR), and Progression-Free Survival (PFS) as assessed by the investigator per RECIST v1.1.
  Overall Survival (OS).
Phase II Study | Approximately 2 years
  Efficacy Endpoints: CBR, DoR, DCR, PFS, and OS as assessed by the investigator per RECIST v1.1.
  Safety Endpoints: Laboratory parameters, 12-lead ECG, echocardiogram, vital signs, physical examination, TEAEs and SAEs.
  Pharmacokinetic Endpoints: Minimum concentration at steady state (Cmin,ss), maximum concentration at steady state (Cmax,ss), degree of fluctuation (DF), average steady-state plasma concentration (Cave,ss), and accumulation index (RAC).

OTHER OUTCOMES:
The sponsor will determine whether and when to conduct exploratory investigations based on the study progress. | Approximately 2 years
  1. Correlation between estrogen receptor (ER) target inhibition, as assessed by 18F-Fluoroestradiol (18F-FES) PET/CT whole-body scans, and treatment efficacy.
  2. FWD1802 metabolic pathway: Identification and concentration measurement of major metabolites of FWD1802 in human plasma (if applicable).
  3. Relationship between the baseline ESR1 mutation types/frequencies and the efficacy of FWD1802. [Time Frame: Approximately 2 years]
  4. Changes in mutation types and frequencies of ESR1 and/or other breast cancer-related biomarkers in ctDNA assays before and after FWD1802 treatment, and the correlation between alterations in the mutational profile and treatment efficacy.(Phase II Study Only)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Principal Investigator — Fudan University
Locations (22):
- China (22):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Huizhou First Hospital, Huizhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - The second people's hospital of Yibin, Yibin, Sichuan
  - Tianjin Medical University Cancer institute & Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital,affiliated with Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT06064812/Prot_000.pdf
  • Informed Consent Form (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT06064812/ICF_001.pdf